CLINICAL TRIAL: NCT04886700
Title: A Single-arm, Open-label, Multicenter, Phase II Study for Evaluation of Efficacy and Safety of the SG001 Injection for Patients With PD-L1-positive Relapsed or Metastatic Uterine Cervical Cancer
Brief Title: Study of the SG001 Injection for Patients With Relapsed or Metastatic Uterine Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSA1802-CSP-004
Record Dates: First submitted 2021-04-26; First posted 2021-05-14 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-05

CONDITIONS: Uterine Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SG001 (Experimental): Recombinant Human Anti-PD-1 Monoclonal Antibody
  Interventions: Drug: SG001

INTERVENTIONS:
Drug: SG001 — Subjects will receive intravenous infusion of SG001 at the dose of 240 mg every 2 weeks until disease progression, unacceptable toxicity, meeting the suspension or termination criteria, or up to 24 months in patients without disease progression.
  Other Names: Recombinant Human Anti-PD-1 Monoclonal Antibody

SUMMARY:
This study is an open, single-arm, multicenter phase II study to investigate the efficacy and safety of SG001 for relapsed or metastatic uterine cervical cancer patients with PD-L1 positive (CPS≧1), and has failed at least first line platinum-based chemotherapy.

DETAILED DESCRIPTION:
Phase II: open, single-arm, multicenter.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 on the day of signing informed consent and volunteered to participated in this study.
* 2. Histologically documented relapsed or metastatic uterine cervical cancer including squamous cell carcinoma, adenocarcinoma, and adenosquamous carcinoma, a relevant pathological report must also be provided.
* 3. Relapsed or metastatic uterine cervical cancer patient who has failed at least first line platinum-based chemotherapy, which means having disease progression during or following at least first line platinum based chemotherapy or for which platinum based chemotherapy is not tolerated, having disease progression within 6 months of or during neoadjuvant or adjuvant treatment with platinum based chemotherapy can also be accepted.
* 4. Programmed Cell Death Ligand 1 (PD-L1) positive expression defined by Combined Positive Score (CPS) ≥1.
* 5. All the subjects should have at least one measurable lesion in CT or MRI test assessed by RECIST 1.1. A previously irradiated site lesion could only be counted as a target lesion if there was clear sign of progression since the irradiation.
* 6. If subjects have received anti-tumor therapies before, the toxicity severity must decrease to ≤ Grade1 evaluated by NCI-CTCAE 5.0, except for residual alopecia or fatigue.
* 7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* 8. Has a predicted survival period ≥ 3 months assessed by investigators.
* 9. Demonstrate adequate organ function as defined below:

  1. Blood routine tests (No blood transfusions were performed, no hematopoietic stimulators were used, and no drugs were used to correct blood cell counts ): Absolute neutrophil count (ANC) ≥1.5×109/L; Platelets ≥75×109/L; Hemoglobin (HGB)≥9 g/dL;
  2. Serum biochemical indexs: Serum creatinine ≤1.5 X ULN or Creatinine clearance (CCr) ≥ 50mL/min; Serum total bilirubin (TBIL) ≤ 1.5 X upper limit of normal ULN (Subjects with Gilbert's syndrome can be up to 3 x ULN); Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 X ULN or ≤5 X ULN for subjects with hepatocellular carcinoma and liver metastases;
  3. Coagulation function: Activated partial thromboplastin time (APPT) and International Normalized Ratio (INR)≤1.5 X ULN (No anticoagulants or other drugs affecting clotting function were used within 14 days prior to the first administration, except for subjects requiring long-term anticoagulant therapy).
* 10. Women of child-bearing potential (WOCBP) should be willing to use reliable contraceptive methods from signing the informed consent form to 6 months after last dose of investigational drug.

Exclusion Criteria:

* 1. History of allergic reactions attributed to any monoclonal antibody, and uncontrolled history of allergic asthma.
* 2. Patients with other types of malignant tumours that have progressed or require treatment within 5 years prior to the screening, but well-treated skin basal cell carcinoma, skin squamous cell carcinoma, or superficial bladder cancer, and having cured carcinoma in situ, e.g. breast carcinoma in situ, can be accepted.
* 3. Patients with any active autoimmune disease, but subjects with following diseases are allowed for further screening: subjects with well-controlled type I diabetes, well-controlled hypothyroidism with hormone replacement therapy, skin diseases (such as vitiligo, psoriasis, or hair loss) without systemic treatment, or who are not expected to relapse without external triggers.
* 4. History of primary immunodeficiency.
* 5. Patients with serious cardiovascular diseases, such as grade 2 or above heart failure based on the NYHA (New York Heart Association) Class guidelines, previous myocardial infarction within 3 months, poorly controlled arrhythmias or unstable angina pectoris, previous arterial or venous thrombosis events within 3 months (e.g. transient ischemic attack, cerebral hemorrhage, cerebral infarction, deep vein thrombosis and pulmonary embolism).
* 6. Has history of Interstitial Lung Disease (Patients caused by radiotherapy are eligible), or non-infectious pneumonitis need for glucocorticoid therapy.
* 7. Have a history of active tuberculosis.
* 8. Subjects with untreated or treated but still symptomatic central nervous system metastases (except for residual signs or symptoms related to CNS treatment, those with stable or improved neurological symptoms at least 2 weeks prior to screening can be included).
* 9. Prior therapy with any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways including anti-PD-1, anti-PD-L1, anti CTLA-4, OX40 agonist, and anti-CD137, etc.
* 10. Immune-related adverse events of grade 3 or higher（NCI-CTCAE 5.0）after immune therapy.
* 11. Have received major surgery or radical radiotherapy within 28 days, or palliative radiotherapy within 14 days, or radiological agents (strontium, samarium, etc.) within 56 days prior to screening.
* 12. Have received systemic anti-tumour therapy 28 days before the first dose, including but not limited to chemotherapy, immunotherapy, macromolecular targeted therapy, and biological therapy (tumour vaccine, cytokines or growth factors controlling cancer); Patients who received small-molecule targeted and oral fluorouracil therapy within 14 days before the first dose.
* 13. Have received attenuated live vaccine within 28 days before the first dose or planned to receive during the study period.
* 14. Have received Chinese herbal medicine or Chinese patent medicine with anti-tumor activity within14 days prior to the first dose.
* 15. Any active infection requiring systemic treatment by intravenous infusion within 28 days prior to the first dose.
* 16. Have received systemic corticosteroids (at doses equivalent to or greater than 10 mg/day of prednisone) or other immunosuppressive drugs within 14 days prior to the first dose of study drug.
* 17. Have participated other clinical trials and received related investigated drugs within 28 days prior to the first dose of study drug (counted from the date of the last treatment in the previous clinical trial, patients participated in the overall survival follow-up of the previous clinical trial can be accepted).
* 18. Patients should be excluded if they have a positive test for human immunodeficiency virus antibody (HIV-Ab) or treponema pallidum antibody (TP-Ab). Patients with positive Hepatitis B virus surface antigen (HBsAg) and/or hepatitis B virus core antibody (HBcAb) as well quantitative HBV-DNA above upper limit of normal value, and patients with positive hepatitis C virus antibody (HCV-Ab) as well quantitative HCV-RNA above upper limit of normal value, should also be excluded.
* 19. Pregnant or lactating women; Or the blood pregnancy test of women at child-bearing age is positive during screening.
* 20. Other conditions that may increase the risk of drug use in the study, or interfere with the interpretation of the study results, or affect the compliance of the study, etc.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 104 (Estimated)
Dates: Start 2021-07-31 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST1.1 in relapsed or metastatic uterine cervical cancer evaluated by IRC (Independent Review Committee), confirmation of CR and PR is required in at least 4 weeks after initial documentation. | From first dose to the first documented progression of disease, subject withdrawal, lose to follow-up, death, initiating a subsequent cancer therapy, or study completion or termination, whichever occurs earliest, assessed up to 24 months.
  To investigate the efficacy of SG001 in relapsed or metastatic uterine cervical cancer.

SECONDARY OUTCOMES:
ORR (objective response rate) evaluated by investigators. | From first dose to the first documented progression of disease, subject withdrawal, lose to follow-up, death, initiating a subsequent cancer therapy, or study completion or termination, whichever occurs earliest, assessed up to 24 months.
  To investigate the efficacy of SG001 in relapsed or metastatic uterine cervical cancer.
DOR (duration of response) evaluated by IRC. | From first dose to the first documented progression of disease, subject withdrawal, lose to follow-up, death, initiating a subsequent cancer therapy, or study completion or termination, whichever occurs earliest, assessed up to 24 months.
  To investigate the efficacy of SG001 in relapsed or metastatic uterine cervical cancer.
DCR (disease control rate) evaluated by IRC. | From first dose to the first documented progression of disease, subject withdrawal, lose to follow-up, death, initiating a subsequent cancer therapy, or study completion or termination, whichever occurs earliest, assessed up to 24 months.
  To investigate the efficacy of SG001 in relapsed or metastatic uterine cervical cancer.
PFS (free-progression survival) evaluated by IRC. | From first dose to the first documented progression of disease, subject withdrawal, lose to follow-up, death, initiating a subsequent cancer therapy, or study completion or termination, whichever occurs earliest, assessed up to 24 months.
  To investigate the efficacy of SG001 in relapsed or metastatic uterine cervical cancer.
OS (overall survival) evaluated by IRC. | From first dose to the first documented progression of disease, subject withdrawal, lose to follow-up, death, initiating a subsequent cancer therapy, or study completion or termination, whichever occurs earliest, assessed up to 24 months.
  To investigate the efficacy of SG001 in relapsed or metastatic uterine cervical cancer.
TTR (time to response) evaluated by IRC. | From first dose to the first documented progression of disease, subject withdrawal, lose to follow-up, death, initiating a subsequent cancer therapy, or study completion or termination, whichever occurs earliest, assessed up to 24 months.
  To investigate the efficacy of SG001 in relapsed or metastatic uterine cervical cancer.
Amount, severity, and duration of TEAEs (treatment emergent adverse event) evaluated by NCI-CTCAE V5.0. | From the date of signing Informed Consent Form (ICF) up to 28 days following the last dose of study drug, immune related adverse events will be recorded until 90 days after the last dose.
  To investigate the safety and tolerance profile of SG001 in patients with relapsed or metastatic uterine cervical cancer.
Population pharmacokinetic parameter IIV (interindividual variability). | At the end of cycle 7 (every cycle is 14 days).
  The pharmacokinetic profile of SG001.
Population pharmacokinetic parameter exposure-response relationship. | At the end of cycle 7 (every cycle is 14 days).
  The pharmacokinetic profile of SG001.
Immunogenicity of SG001, such as anti-drug antibody and neutralizing antibody. | From the first dose of study drug to the end of treatment visit, up to 24 months.
  To investigate the immune profile of SG001.

CONTACTS AND LOCATIONS:
Overall Officials: Lingying Wu, Medical PhD, Principal Investigator — Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- National Cancer Center/Cancer Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li G, Li X, Yin R, Feng M, Zuo J, Wei S, Kang S, Sun H, Li X, Wang Y, Zhang Y, Sun L, Lin D, Ruan X, Zhu Z, Jiang K, Liu H, Wang W, Hao D, Chen Y, Xiang S, Niu M, Wu L. Phase II study of enlonstobart (SG001), a novel PD-1 inhibitor in patients with PD-L1 positive recurrent/metastatic cervical cancer. Gynecol Oncol. 2024 Dec;191:165-171. doi: 10.1016/j.ygyno.2024.10.001. Epub 2024 Oct 23. PMID 39447517